CLINICAL TRIAL: NCT03977909
Title: Early Maladaptative Schemas Among Euthymic Patients With Bipolar Disorder: Exploring the Relationships With Symptoms, Functioning and Cognition in the Versailles FondaMental Advanced Centers of Expertise for Bipolar Disorders
Brief Title: Early Maladaptative Schemas Among Euthymic Patients With Bipolar Disorder in the Versailles FondaMental Advanced Centers of Expertise for Bipolar Disorders Cohort
Acronym: SPIBIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Collaborators: Fondation FondaMental (Other); Versailles Saint-Quentin-en-Yvelines University (Other); University of Bordeaux (Other)
Responsible Party: Principal Investigator, Dr Paul ROUX, Psychiatre, Maître de Conférence des Université Praticien Hospitalier, Versailles Hospital
Other Study IDs: CHVersailles
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Bipolar Disorder
Keywords: Early Maladaptative Schemas; Cognition; Functioning
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early Maladaptive Schemas (EMS) are overactivated in euthymic bipolar disorders (BD) and are associated with poor psychosocial functioning and higher suicidality.

The first objective of this study is to establish different clusters of EMS in euthymic bipolar disorders, compare these clusters according to the clinical characteristics of BD and neuropsychological performances and evaluate the temporal stability of these clusters at 12 and 24 months.

The second objective of this study is to quantify the impact of EMS on functioning in euthymic BD, beyond the effect of cognition and residual depressive symptoms.

DETAILED DESCRIPTION:
Early Maladaptive Schemas (EMS) are overactivated in euthymic bipolar disorders (BD) and are associated with poor psychosocial functioning and higher suicidality. However, few studies have explored EMS in bipolar disorders, despite EMS therapy is a promising tool for the psychotherapy of BD.

This study will use the data collected at the Versailles Expert Center for Bipolar disorder, in the local FACE-BD registry. These data will be collected at the inclusion, 12 months and 24 months later. They included an extensive neuropsychological battery and an extensive evaluation of the clinical characteristics of bipolar disorder. EMS will be measured with the Young Schema Questionnaire Short Form 3.

The first objective of this study is to establish different clusters of EMS in euthymic bipolar disorders, compare these clusters according to the clinical characteristics of BD and neuropsychological performances and evaluate the temporal stability of these clusters at 12 and 24 months.

The second objective of this study is to quantify the impact of EMS on functioning in euthymic BD, beyond the effect of cognition and residual depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

- bipolar disorder according to DSM IV-R (structured clinical interview)

Exclusion Criteria:

* major depressive or manic or hypomanic during the evaluation
* Montgomery Åsberg Depression Rating Scale ⩽10
* Young Mania Rating Scale ⩽12

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients recruited into the FACE-BD (FondaMental Advanced Centers of Expertise for Bipolar Disorders) cohort at Versailles Hospital. This registry was set up by the Fondation FondaMental (www.fondation-fondamental. org) which created an infrastructure and provided resources to follow clinical cohorts and comparative-effectiveness research in patients with BD.
  Patients were referred by their general practitioner or by their psychiatrist.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Early Maladaptative Schemas T0 | 18 measures by subject, assessed at inclusion
  distance to the norm for the scores on each 18 early maladaptative schema measured with the Young Shema Questionnaire short form 3, no lower bound limit, no upper bound limit, a low score indicate a lower activation of the Early Maladaptative Schema
Early Maladaptative Schemas T12 | 18 measures by subject, assessed at 12 months
  distance to the norm for the scores on each 18 early maladaptative schema measured with the Young Shema Questionnaire short form 3, no lower bound limit, no upper bound limit, a low score indicate a lower activation of the Early Maladaptative Schema
Early Maladaptative Schemas T24 | 18 measures by subject, assessed at inclusion 24 months
  distance to the norm for the scores on each 18 early maladaptative schema measured with the Young Shema Questionnaire short form 3, no lower bound limit, no upper bound limit, a low score indicate a lower activation of the Early Maladaptative Schema

SECONDARY OUTCOMES:
functioning | one measure by subject, assessed 3 times (inclusion, 12 months and 24 months)
  total score on the Functioning Assessment Short Test (lower bound 0 upper bound 72, lower scores indicates better functioning)
Depression | one measure by subject, assessed 3 times (inclusion, 12 months and 24 months)
  total score on the Montgomery Åsberg Depression Rating Scale (minimum 0 maximum 10)
Cognition | 5 measures by subject, assessed 2 times (at inclusion and 24 months)
  distance to the norm for the scores for each the five cognitive dimension measured with the standardised neuropsychological battery, no lower bound limit, no upper bound limit, lower scores indicate poorer cognition
Hypomania | one measure by subject, assessed 3 times (inclusion, 12 months and 24 months)
  total score on the Young Mania Rating Scale (lower bound 0 upper bound 12, lower scores indicate lower hypomania

CONTACTS AND LOCATIONS:
Locations (1):
- Paul ROUX, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball J, Mitchell P, Malhi G, Skillecorn A, Smith M. Schema-focused cognitive therapy for bipolar disorder: reducing vulnerability to relapse through attitudinal change. Aust N Z J Psychiatry. 2003 Feb;37(1):41-8. doi: 10.1046/j.1440-1614.2003.01098.x. PMID 12534655
- [Background] Hawke LD, Provencher MD, Parikh SV. Schema therapy for bipolar disorder: a conceptual model and future directions. J Affect Disord. 2013 May 15;148(1):118-22. doi: 10.1016/j.jad.2012.10.034. Epub 2012 Dec 4. PMID 23218898
- [Background] Morriss R. Clinical importance of inter-episode symptoms in patients with bipolar affective disorder. J Affect Disord. 2002 Dec;72 Suppl 1:S3-13. doi: 10.1016/s0165-0327(02)00340-3. PMID 12589898
- [Background] Nilsson KK. Early maladaptive schemas and functional impairment in remitted bipolar disorder patients. J Behav Ther Exp Psychiatry. 2012 Dec;43(4):1104-8. doi: 10.1016/j.jbtep.2012.05.005. Epub 2012 Jun 7. PMID 22743343
- [Background] Roux P, Raust A, Cannavo AS, Aubin V, Aouizerate B, Azorin JM, Bellivier F, Belzeaux R, Bougerol T, Cussac I, Courtet P, Etain B, Gard S, Job S, Kahn JP, Leboyer M, Olie E; FondaMental Advanced Centers of Expertise in Bipolar Disorders (FACE-BD) Collaborators; Henry C, Passerieux C. Associations between residual depressive symptoms, cognition, and functioning in patients with euthymic bipolar disorder: results from the FACE-BD cohort. Br J Psychiatry. 2017 Dec;211(6):381-387. doi: 10.1192/bjp.bp.117.201335. Epub 2017 Oct 19. PMID 29051175
- [Background] Urosevic S, Abramson LY, Harmon-Jones E, Alloy LB. Dysregulation of the behavioral approach system (BAS) in bipolar spectrum disorders: review of theory and evidence. Clin Psychol Rev. 2008 Oct;28(7):1188-205. doi: 10.1016/j.cpr.2008.04.004. Epub 2008 May 9. PMID 18565633
- [Background] Young, J. E., & Brown, G. (1998). Young schema questionnaire short form. New York: Cognitive Therapy Center.
- [Background] Young, J. E., Klosko, J. S., & Weishaar, M. E. (2003). Schema therapy: A practitioner's guide, Guilford Press.